CLINICAL TRIAL: NCT04427228
Title: MIGRAINE: Randomized trIal of Single Versus Multifraction Radiosurgery on Immunotherapy
Brief Title: Single vs Multi-fraction SRS Patients on Immunotherapy
Acronym: MIGRAINE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB19-2022
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Brain Cancer; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Radiation: Radiosurgery Three Treatments
- ARM B (Active Comparator)
  Interventions: Radiation: Radiosurgery Single Treatment

INTERVENTIONS:
Radiation: Radiosurgery Single Treatment — Frameless single-fraction SRS. One large treatment done on each brain tumor. 20 Gy for GTVs (or resection cavity CTVs) < 2 cm, and 18 Gy for GTVs (or resection cavity CTVs) between 2-3 cm in the single-fraction.
  Other Names: SRS
  Arms: ARM B
Radiation: Radiosurgery Three Treatments — Multi-fraction SRS. Three small doses done on each brain tumor. 27 Gy in 3 fractions in the multi-fraction group
  Other Names: SRS
  Arms: Arm A

SUMMARY:
This study is meant to compare different surgical approaches to brain cancer.

ELIGIBILITY:
Inclusion Criteria:

i. Adult patients (≥ 18 years old) with an ECOG Performance Status 0-2 and a life expectancy of 3 months or more.

ii. Histologically confirmed systemic malignancy with gadolinium contrast-enhanced MRI scan demonstrating 1-10 newly diagnosed intraparenchymal brain metastases.

iii. Well-circumscribed, measureable intraparenchymal brain metastasis(s) with maximum tumor diameter ≤3.0 cm. If multiple metastases are present, the other(s) must not exceed 3.0 cm in maximum diameter. At least one metastasis must be ≥ 0.5 cm in maximum diameter to be considered measurable disease.

iv. Negative urine or serum pregnancy test done ≤ 21 days prior to CT simulation, for women of child bearing potential only.

v. Ability to understand and willingness to sign a written informed consent document.

vi. Must have received immunotherapy (PD-1/PD-L1 and/or CTLA-4 inhibitor(s)) within the past 6 months or plan on receiving immunotherapy within the next 1 month.

vii. Must have a Gustave Roussy Immune Score (GRIm-Score) of 0 or 1 (neutrophil-to-lymphocyte ratio > 6 = 1 point, LDH > Upper Limit of Normal = 1 point, and Albumin < 3.5 g/dL = 1 point).

Exclusion Criteria:

i. Diagnosis of germ cell tumor or hematologic malignancy. ii. Metastases in the brain stem, midbrain, pons, medulla, or within 7 mm of the optic apparatus (optic nerves, chiasm and optic tracts).

iii. Diagnosis of leptomeningeal disease. iv. Prior SRS to an immediately adjacent lesion(s) of interest or to the current lesion(s) of interest.

v. Prior history of pseudoprogression or radionecrosis from cranial radiotherapy.

vi. A neurosurgical resection cavity deemed too large by the radiation oncologist to be treated with a single fraction of stereotactic radiosurgery.

vii. Contraindications to gadolinium contrast-enhanced MRI (eg, non-compatible pacemaker, eGFR <30, gadolinium allergy).

viii. A Gustave Roussy Immune Score (GRIm-Score) > 1 (neutrophil-to-lymphocyte ratio > 6 = 1 point, LDH > Upper Limit of Normal = 1 point, and Albumin < 3.5 g/dL = 1 point).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Multi-Fraction SRS superiority compared to single fraction SRS | 4 years
  To determine if Multi-Fraction SRS will decrease the rate of radionecrosis when compared to single-fraction SRS for patients with small metastases and are on immunotherapy.

SECONDARY OUTCOMES:
Target metastasis progression | 4 years
  Target metastasis progression will be assessed using adapted Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) consensus imaging criteria. In brief, progressive disease is defined as a ≥20% relative increase in the longest diameter (LD) of the target metastasis compared to its smallest LD recorded on study, with a minimum absolute increase of 5 mm
Overall Survival Rate | 4 years
  Time from randomization to death
Acute CTCAE v5.0 CNS Grade 2+ and Grade 3+ toxicities | 4 years
  Any acute CTCAE v5.0 CNS Grade 2+ and Grade 3+ toxicities, within 90 days of SRS completion (toxicity must be specified).
Late CTCAE v5.0 CNS Grade 2+ and Grade 3+ toxicities | 4 years
  Any late CTCAE v5.0 CNS Grade 2+ and Grade 3+ toxicities, greater than 90 days from SRS completion (toxicity must be specified).
rate of individual metastases radionecrosis | 4 years
  To compare the rates over time of individual metastases radionecrosis using a parametric survival analysis
rate of individual metastases rates of edema | 4 years
  To compare rates over time of individual metastases rates of edema using a parametric survival analysis.
Rates of Symptomatic Edema | 1 year
  To compare rates of symptomatic edema at 3 months, 6 months, and 1 year.1
Time to any distant intracranial failure | 4 years
  Time to any distant intracranial failure (ie, appearance of brain metastasis at untreated site).
Time to initiation of any combination | 4 years
  Time to initiation of any combination of death, salvage SRS, WBRT, or neurosurgical resection for intracranial failure.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago, Chicago, Illinois, United States